CLINICAL TRIAL: NCT05370014
Title: Improving the Collaborative Health of Minority COVID-19 Survivor and Carepartner Dyads Through Interventions Targeting Social and Structural Health Inequities.
Brief Title: Improving the Collaborative Health of Minority COVID-19 Survivor and Carepartner Dyads
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Gayenell S. Magwood, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00110062; 1R01NR020127-01 (NIH)
Record Dates: First submitted 2022-04-14; First posted 2022-05-11 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: SARS- CoV-2; Cardiovascular Diseases; Chronic Kidney Diseases; Diabetes Mellitus, Type 2; Chronic Disease; Stroke
Keywords: health inequities; rural; Black/African American; dyads; structural determinants of health; quality of life
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Chronic Disease; Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCINGS Fam Intervention (Experimental): Integrating Community-based Intervention Under Nurse Guidance with Families (iCINGS FAM) is 14-week, nurse coordinated, Community Health Worker (CHW) supported telehealth intervention structure. After baseline assessment, dyads randomized to the intervention group (n= 125 dyads) will have two planning sessions (over 2 weeks) followed by eight topic-guided sessions delivered by a member of the RN-CHW team over 12 weeks (weekly the first 4 weeks, then bi-weekly), Follow up assessments will occur at month 4 and month 7.
  Interventions: Behavioral: Integrating Community-based Intervention Under Nurse Guidance with Families (iCINGS FAM)
- Attention Control (No Intervention): After baseline assessment, dyads randomized to the attention control group (n= 125 dyads) will receive monthly (3 in total; 7-10 min each) scripted phone calls on focused on general health risks and health promotion. Monthly telephone calls will cover readily accessible evidence-based public health messaging from the Centers for Disease Control and Prevention (CDC) Your Health, NIH and other public health community facing websites related to COVID-19 mitigation such as risk reduction and prevention strategies including flu vaccines, asymptomatic spread, and contact tracing. Follow up assessments will occur at month 4 and month 7.

INTERVENTIONS:
Behavioral: Integrating Community-based Intervention Under Nurse Guidance with Families (iCINGS FAM) — The intervention consists of two planning sessions with the dyad (over 2 weeks) followed by eight topic-guided sessions delivered the RN-CHW team over 12 weeks (weekly the first 4 weeks, then bi-weekly) (Table 3). Key components of these televisits include COVID-19 risk mitigation, chronic disease management, medication adherence, family functioning/support, and community and health systems resource identification and referral with ongoing goal planning. The RN-CHW will meet weekly for progress review, follow up planning, and setting up anticipatory guidance for the next session with the dyads. The RN and CHW will also review IC or survivor dissatisfaction and other issues that require more immediate attention. RN-CHW planning will be assessed to make sure each televisit remain topic focused yet incorporates flexibility to suit the needs of each dyad.
  Arms: iCINGS Fam Intervention

SUMMARY:
This study tests the efficacy of a dyadic intervention to mitigate the adverse health consequences of severe acute respiratory syndrome coronavirus 2 (SARS- CoV-2 )(COVID-19) in African American (AA) adults with pre-existing chronic health conditions and their informal carepartners (IC). Socioeconomically disadvantaged, older, and Black/African American from rural regions are burdened with greater rates of chronic diseases such as diabetes, hypertension, chronic kidney disease, cardiovascular disease, and stroke.

DETAILED DESCRIPTION:
This study tests the efficacy of a dyadic intervention to mitigate the adverse health consequences of SARS- CoV-2 (COVID-19) in African American (AA) adults with pre-existing chronic health conditions and their informal carepartners (IC). Socioeconomically disadvantaged, older, and Black/African American from rural regions are burdened with greater rates of chronic diseases such as diabetes, hypertension, chronic kidney disease, cardiovascular disease, and stroke. Those chronic diseases contribute to more severe health consequences and higher rates of mortality from COVID-19. POC are also more likely to be impacted by social and structural determinants of health (SSDH), such as barriers to health care access, discrimination, and lack of social support, that negatively impact quality of life (QoL) and effective chronic disease self- management behaviors. To provide the fullest health benefits to participants with chronic conditions in the wake of the COVID-19 pandemic, it is critical that we design interventions targeting SSDH for improved chronic disease self-management, health, functioning, QoL.

This study will utilize an embedded mixed methods design paired with an efficacy randomized controlled trial (RCT). Our iCINGS FAM (Integrating Community-based Intervention Under Nurse Guidance with Families) is a Registered Nurse (RN)-Community Health Worker (CHW)-delivered, telehealth intervention (14-weeks) that targets compounding racial- and pandemic-related stressors for improved chronic illness management and future disease risk mitigation in adult AA COVID-19 survivor/IC dyads.

ELIGIBILITY:
Inclusion Criteria:

COVID-19 survivor inclusion criteria

* African American
* Male and female
* Living in a Medically Underserved Area and/or a designated rural area of South Carolina
* ≥ 18 years and above
* A history of a COVID-19-associated hospitalization, ER or Urgent Care visit since March 11th, 2020
* A previous diagnosis of one or more of the following conditions: type 2 diabetes, hypertension, cardiovascular disease, chronic kidney disease, or stroke (>3 months)

  -Carepartner inclusion criteria
* Male and female
* ≥ 18 years and above
* Must live on the same property or community, preferably within a 40-mile radius of the survivor
* Primarily responsible for care provision and/or care/social support in the home (i.e., is not paid for services)

Exclusion Criteria:

* Survivor and Carepartner exclusion criteria • Enrolled in related clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported outcomes measurement information system (PROMIS) Global Health Scale | 0, 4, 7 months
  Quality of Life 10 items. minimum score 4 to maximum score 20. Higher scores mean better.

SECONDARY OUTCOMES:
Change in PROMIS Short Form v1.0 Anxiety | 0, 4, 7 months. minimum score 6 to maximum score 30. lower scores mean better.
  Anxiety 6a (6 items)
Change in Center for Epidemiologic Studies Depression Scale (CES-D) | 0, 4, 7 months
  Depression 20 items. minimum score 0 to maximum score 60. lower scores mean better.
Change in PROMIS Short Form v1.0 Fatigue | 0, 4, 7 months
  Fatigue 6a (6 items). minimum score 6 to maximum score 30. lower scores mean better.
Change in PROMIS Short From v1.0 Sleep Disturbance | 0, 4, 7 months
  Sleep Disturbance 6a (6 items). minimum score 6 to maximum score 30. lower scores mean better.
Change in PROMIS Short Form v.1.1 Pain interference | 0, 4, 7 months
  Pain interference 8a (8 items). minimum score 8 to maximum score 40. lower scores mean better.
Change in Dyadic Illness Management Behaviors | 0, 4, 7 months
  Survivor reported Self-care chronic illness Inventory (20 items); Informal carepartner contributions to self-care of chronic illness inventory 20 item
Change in Dyadic Efficacy | 0, 4, 7 months. minimum score 10 to maximum score 50. higher scores mean better.
  PROMIS v1.0 General Self-efficacy Scale (10 items)
Change in Modified Medical Outcomes Study Social Support Survey Instrument (mMOS-SS) | 0, 4, 7 months
  Social Support (8 items). Transformed minimum score 0 to maximum score 100. higher scores mean better.

CONTACTS AND LOCATIONS:
Overall Officials: Gayenell S Magwood, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott J, Burrison S, Barron M, Logan A, Magwood GS. Exploring Nursing Strategies to Engage Community in Cardiovascular Care. Curr Cardiol Rep. 2023 Oct;25(10):1351-1359. doi: 10.1007/s11886-023-01949-9. Epub 2023 Sep 4. PMID 37665520
- [Result] Magwood GS, Ellis C Jr, Hughes Halbert C, Toussaint EA, Scott J, Nemeth LS. Exploring Barriers to Effective COVID-19 Risk Mitigation, Recovery, and Chronic Disease Self-Management: A Qualitative Multilevel Perspective. Patient Relat Outcome Meas. 2024 Sep 18;15:241-253. doi: 10.2147/PROM.S467743. eCollection 2024. PMID 39310085